CLINICAL TRIAL: NCT04553536
Title: Perioperative Cardiovascular Protection Conservative Effects of Esketamine Versus µ-opioid Receptor Agonists in Total Intravenous General Anesthesia: Study Protocol for a Randomized Controlled Pilot Trial
Brief Title: Cardiovascular Protection Conservative Effects of Esketamine Versus µ-opioid Receptor Agonists in General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZGuo20200826
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Opioid Analgesic Adverse Reaction
MeSH Terms: interventions — Esketamine; Propofol; Atracurium; cisatracurium; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid analgesics (Active Comparator): Mu-opioid receptor agonists (remifentanil, sulfentanil) will be used as the only analgesic(s) in the surgery.
  Interventions: Drug: Esketamine, Sulfentanil or/and Remifentanil
- Ketamine (Experimental): Esketamine will be used as the only anagesic in the surgey.
  Interventions: Drug: Esketamine, Sulfentanil or/and Remifentanil

INTERVENTIONS:
Drug: Esketamine, Sulfentanil or/and Remifentanil — The esketamine or the opioids will be intravenously injected or infused to the patients with propofol and one of the muscle relaxants to induce and maitain general anesthesia.
  Other Names: Propofol, Atracurium Besilate or Cisatracurium besylate or Rocuronium Bromide

SUMMARY:
Pain is 'a double-edged sword', disturbing daily life of the sufferers and activating the intrinsic protective mechanisms. Transient receptor potential vanilloid 1 (TRPV1), play such role as 'a double agent', transmitting the pain signals and initiating the cardio-protective mechanism via release protective neuropeptides.

Surgery-related pain is mostly so severe and disturbing that must be medically treated. Unfortunately, the beneficial aspect of pain is commonly ignored in daily clinical practice. Does it matter to the patients' outcomes? We don't know yet! What we have been seeing is the shocking outcomes of patients underwent surgery, which shows about 0.8% and 7% of mortalities in the period of 48 hours and 30 days after surgery, respectively (https://www.rcplondon.ac.uk/projects/outputs/national-hip-fracture-database-annual-report-2016; Injury. 2017; 48(10): 2180-2183). What causes the disaster? Piles of evidence demonstrate that deep anesthesia or deep sedation is related to the high mortality of the patients (Anesthesiology. 2012; 116:1195-1203; Crit Care. 2014; 18(4):R156 ). What about the effect of analgesia, especially the over-analgesia, on the patients' outcome in and after surgery? Opioids are the most commonly used drugs in the treatment of moderate and sever pain including intra- and postoperative pain. The µ-opioid receptor agonists induce analgesic effect via inhibition of the transduction and the transmission of pain signals, by suppression of the release of CGRP and SP from the nerve terminals. The protective effects on cardiovascular system mediated by CGRP and SP can be inhibited, if the same effect is produced by the action of opioids in the peripheral nerve terminals innervating the heart and the vasculature. Our previous research shows that intrathecal administration of morphine or epidural administration of ropivacaine (1%, in 20 μL) significantly attenuates the increases of CGRP and its coding mRNA in ventricular myocardium and the innervating dorsal root ganglion neurons following occlusion of coronary artery in experimental animals. We design this study to investigate the potential adverse effect of anesthesia with opioid as the main analgesic.

DETAILED DESCRIPTION:
We hypothesize that over-analgesia using opioids significantly suppresses the activity of TRPV1/CGRP and SP and reduces the amount of CGRP and SP released, which results in an effective de-protection of the cardiovascular system. The severer myocardial damage under some insulting circumstances and eventful systemic hemodynamics is likely occurring upon some surgical/pathological/pharmacological insults in the intra- and postoperative periods.

This parallel, randomized controlled trial will be conducted in eleven centers in Shanxi province, China, which is designed to investigate the perioperative incidence of adverse cardiovascular events and alteration of cardiac troponin I (cTnI) in the patients (one thousand patients, ASA Physical Status 1-II, older than 16 years, regardless of the gender) undergoing surgery under total intravenous general anesthesia with conventional µ-opioid agonists or Esketamine, as the major analgesic. Clinically appropriate anesthesia depth or BIS readings will be used for judgement of anesthetic depth. Conventional monitoring parameters, including blood pressures, heart rate, SpO2 and ECG, will be recorded and analyzed. Blood samples will be collected at 30 min before induction of anesthesia, at the end of surgery and 24 h after the surgery. The association of the perioperative adverse cardiovascular events and the alterations of the levels of serum TRPV1, CGRP, SP and cTnI in the patients underwent general anesthesia using different analgesics (µ-opioid agonists vs Esketamine) will be evaluated. Postoperative outcome, including the functions of the brain and cardiovascular system, is also going to be traced for 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia

Exclusion Criteria:

* Patients with diabetes and neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative adverse cardiac events | 72 hours
  It includes intra- and post-operative adverse cardiac events.
Cardiac protection related molecules, including transient receptor potential vanilloid 1 (TRPV1), calcitonin gene-related peptide (CGRP) and substance P. | 24 hours
  The molecules exist in myocardium participating in carioprotection.

CONTACTS AND LOCATIONS:
Locations (1):
- Zheng Guo, Taiyuan, Shanxi, China